CLINICAL TRIAL: NCT02974400
Title: Evaluation of Internet-based Cognitive Behavioral Self-help Treatments for Persecutory Ideation and Auditory Verbal Hallucinations
Brief Title: Evaluation of Internet-based Cognitive Behavioral Self-help Treatments for People With Psychosis
Acronym: EviBaS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 159384
Record Dates: First submitted 2016-11-16; First posted 2016-11-28 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Schizophrenia; Hallucinations; Persecutory Delusion
Keywords: internet-based intervention; e-mental health; cognitive behavioural intervention
MeSH Terms: conditions — Schizophrenia; Hallucinations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based guided self-help (Experimental): Internet-based, guided, CBT-oriented self-help treatment for persecutory ideation and auditory verbal hallucinations with access to a self-help website including regular written electronic contact with a guide and access to smartphone-based interactive worksheets (8 weeks)
  Interventions: Behavioral: Internet-based, CBT-oriented, guided self-help
- Wait-List (No Intervention): Wait-list control group (8 weeks)

INTERVENTIONS:
Behavioral: Internet-based, CBT-oriented, guided self-help — The self-help program includes sessions regarding (1) cognitive model, (2) sleep hygiene, (3) mindfulness, (4) meta-cognition, (5) coping with voice hearing, (6) persecutory ideation, (7) worrying, (8) self-esteem, (9) depression, (10) social competence, and (11) relapse prevention.
  Arms: Internet-based guided self-help

SUMMARY:
Schizophrenia is a severe mental disorder which is accompanied by an enormous individual and societal burden. Despite established efficacy of cognitive behavioral therapy for psychosis (CBTp), its dissemination into routine mental health care remains poor. National regulations such as the National Institute for Health and Care Excellence (NICE) guideline in the United Kingdom recommend that CBTp should be offered to every person with psychotic symptoms, but more than 50% do not receive even a single session of CBTp. In Germany, CBTp is virtually not represented in the psychotherapy health service. Internet-based cognitive behavioral therapy (CBT) in a self-help format has been proven feasible and effective in anxiety and depressive disorders. Recently, Internet-based (self-help) interventions are also deployed via smartphone apps. The feasibility of Internet-based treatments for people with schizophrenia is well documented for Internet-based interventions (e.g., medication management) and also reported for smartphone interventions. However, there is a dearth of empirical studies precluding a conclusive picture. As far as the investigators know, there is only one study encompassing 90 participants with psychosis that investigated an Internet-based intervention with symptom-specific, cognitive behavioral interventions, which is from the investigators' research group. The unique features of the proposed project are 1) the first-time evaluation of a symptom-oriented, CBTp-based self-help treatment for people with psychotic symptoms via Internet, enhanced with smartphone assistance. The study is set up as randomized controlled trial (RCT) with active treatment versus a wait-list control group. It evaluates a combined Internet-based guided self-help treatment for persecutory ideation and auditory verbal hallucinations. The active treatment condition consists of access to a self-help website including regular written electronic contact with a guide and access to smartphone-based interactive worksheets (apps). The trials combine the low-threshold advantages of an online approach (e.g., anonymity) with the virtues of a clinical trial (e.g., symptom assessment and diagnostic verification via Interview). The primary outcome measure is the Positive and Negative Syndrome Scale (PANSS). Secondary outcome measures include self-reported symptom measures (Paranoia Checklist; Beliefs About Voices Questionnaire revised), completion rates, drop-out from the intervention, general symptomatology, side-effects, and client satisfaction. The project will help to answer the empirical question whether CBTp-based interventions in a purely Internet-based self-help format are effective. Positive findings would pave the way for an easy-to-access treatment option for patients with psychotic symptoms who currently are deprived of psychotherapeutic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Electronic informed consent
* Internet access
* Adequate command of the German language
* PANSS Suspiciousness/persecution >= 3 AND/OR PANSS hallucinations >=3
* Diagnosis of schizophrenia, schizoaffective disorder or delusional disorder
* Concurrent psychopharmacological treatment

Exclusion Criteria:

* Acute suicidality
* Acute risk of endangering others
* No emergency plan (with is formulated during the telephone interview)
* Disease of the central nervous system with need for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Change in PANSS from pre-intervention to post-intervention (i.e. between 1 and 7 days after completion of the last module)
  Kay et al. (1987); clinician administered

SECONDARY OUTCOMES:
Paranoia Checklist (PC) | Change in PC from pre-intervention to post-intervention (i.e. between 1 and 7 days after completion of the last module)
  Freeman et al. (2005); self-report
Launay-Slade Hallucination Scale (LSHS) | Change in LSHS from pre-intervention to post-intervention (i.e. between 1 and 7 days after completion of the last module)
  Bentall & Slade (1985); self-report
Patient Health Questionnaire (PHQ-9) | Change in PHQ-9 from pre-intervention to post-intervention (i.e. between 1 and 7 days after completion of the last module)
  Spitzer, Kroenke & Williams, 1999; self-report
Incongruence Scale (INK) | Change in INK from pre-intervention to post-intervention (i.e. between 1 and 7 days after completion of the last module)
  Grosse Holtforth, Grawe & Tamcan (2004); self-report
Quality of life (WHO-QOL) | Change in WHO-QOL from pre-intervention to post-intervention (i.e. between 1 and 7 days after completion of the last module)
  WHO; self-report

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Westermann, Dr, Principal Investigator — University of Bern; Steffen Moritz, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (2):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- University of Bern, Bern, Switzerland

REFERENCES:
- [Derived] Westermann S, Ruegg N, Ludtke T, Moritz S, Berger T. Internet-based self-help for psychosis: Findings from a randomized controlled trial. J Consult Clin Psychol. 2020 Oct;88(10):937-950. doi: 10.1037/ccp0000602. Epub 2020 Aug 13. PMID 32790453
- [Derived] Ludtke T, Platow-Kohlschein H, Ruegg N, Berger T, Moritz S, Westermann S. Mindfulness Mediates the Effect of a Psychological Online Intervention for Psychosis on Self-Reported Hallucinations: A Secondary Analysis of Voice Hearers From the EviBaS Trial. Front Psychiatry. 2020 Apr 3;11:228. doi: 10.3389/fpsyt.2020.00228. eCollection 2020. PMID 32308631
- [Derived] Ruegg N, Moritz S, Berger T, Ludtke T, Westermann S. An internet-based intervention for people with psychosis (EviBaS): study protocol for a randomized controlled trial. BMC Psychiatry. 2018 Apr 13;18(1):102. doi: 10.1186/s12888-018-1644-8. PMID 29653532